CLINICAL TRIAL: NCT04613232
Title: Feasibility of Monitoring Patients During Radiotherapy Using Biometric Sensor Data: the OncoWatch Study 1.0
Acronym: OncoWatch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Helle Pappot, Professor, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OncoWatch 1.0
Record Dates: First submitted 2020-10-21; First posted 2020-11-03 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Head and Neck Cancer
Keywords: Smartwatch; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apple Watch (Experimental): The research intervention is continuously monitoring of heart rate and physical activity (minimum 12h/day) with a smartwatch which is connected to a smartphone.
  Interventions: Device: Wearable sensor

INTERVENTIONS:
Device: Wearable sensor — The patients will be asked to wear an Apple Watch during their treatment course. The watch will pasively collect sensor data (heart rate and physical activity)
  Other Names: Smartwatch; Apple watch

SUMMARY:
The aim of the study is to determine the adherence to using an Apple Watch during curative intended radiotherapy for head and neck cancer. Secondly it will bring new insights to the patient's activity levels and how heart rate varies during treatment course.

DETAILED DESCRIPTION:
Patients with head and neck cancer (HNC) experience severe side effects during radiotherapy (RT). Ongoing technological advances in wearable biometric sensors allow for real-time collection of objective data e.g. physical activity and heart rate, which in the future might help to detect and act against side effects before they become severe. A smartwatch such as the Apple Watch allows for objective data monitoring outside hospital with minimal effort for the patient. To find out if such tools can be implemented in the oncological setting feasibility studies are needed.

The aim of the study is to determine the adherence to using an Apple Watch during curative intended radiotherapy for head and neck cancer. Secondly it will bring new insights to the patient's activity levels and how heart rate varies during treatment course.

The study will assess the feasibility of using the Apple Watch for home monitoring of patients with HNC. It will bring new insights to the patient's activity levels and how heart rate varies during treatment course. This is important knowledge before further investigating how biometric data can be used as part of symptom monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Danish patients ≥18 years planned to primary or post-operative curative radiotherapy for squamous-cell carcinoma of the head and neck at Rigshospitalet, University Hospital, Department of Oncology, Denmark.
* Able to read and speak Danish

Exclusion Criteria:

* Seious cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who could wear the device more than 12 hours per day | 3 months
  To determine the feasibility of using an Apple Watch to obtain biometric data for patients undergoing head and neck locoregional therapy throughout the duration of radiotherapy

SECONDARY OUTCOMES:
Data acquisition rate | 3 months
  Percentage of successful data acquisition events

OTHER OUTCOMES:
Change in heart rate | 3 months
  Description of change in hear rate during radiotherapy
Change in physical activity (steps per day) | 3 months
  Description of change insteps per day during radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Holländer-Mieritz, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hollander-Mieritz C, Vogelius IR, Kristensen CA, Green A, Rindum JL, Pappot H. Using Biometric Sensor Data to Monitor Cancer Patients During Radiotherapy: Protocol for the OncoWatch Feasibility Study. JMIR Res Protoc. 2021 May 13;10(5):e26096. doi: 10.2196/26096. PMID 33983123